CLINICAL TRIAL: NCT06781918
Title: BRAIN DEVELOPMENT, GROWTH and HEALTH in CHILDREN with SEVERE ACUTE MALNUTRITION
Brief Title: Severe Acute Malnutrition and Child Development Clinical Trial in Mwanza
Acronym: BRIGHTSAM
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Collaborators: University of Liverpool (Other); Bugando Medical Centre (Unknown); University of Turku (Other); Rigshospitalet, Denmark (Other); University of Copenhagen (Other); Sokoine University of Agriculture (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Dr George PrayGod, Chief Research Scientist, National Institute for Medical Research, Tanzania
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DFC file no. 23-13-RH; DFC file no. 23-13-RH (Other Grant/Funding Number: DANIDA under Danish Ministry of Foreign Affairs)
Record Dates: First submitted 2024-12-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Severe Acute Malnutrition in Childhood
Keywords: Severe acute malnutrition; Ready to use therapeutic food; Childhood development; Psychosocial stimulation; Choline; Docosahexaenoic acid (DHA)
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Intervention Model Description: This is a 2x2 factorial randomized clinical trial which aims to study the effects of DHA and choline enriched ready to use therapeutic foods and psychosocial stimulation in the management of children with severe acute malnutrition.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- eRUTF (Experimental): Choline and DHA enriched Ready to use therapeutic foods
  Interventions: Dietary Supplement: Ready to Use Therapeutic Food (RUTF)
- sRUTF (Placebo Comparator): Standard ready-to-use therapeutic foods
  Interventions: Dietary Supplement: Ready to Use Therapeutic Food (RUTF)
- PS (Experimental): Psychosocial stimulation
  Interventions: Behavioral: Psychosocial stimulation
- sNC (Placebo Comparator): Standard nutritional counseling and psychosocial stimualtion
  Interventions: Behavioral: Psychosocial stimulation

INTERVENTIONS:
Dietary Supplement: Ready to Use Therapeutic Food (RUTF) — DHA & Choline enriched RUTF The modified RUTF is a peanut butter paste that contains vegetable oil, skim milk powder, carbohydrates, vitamins, and minerals the same nutrients which are the same as the standard RUTF but is fortified additionally with 250 mg of choline and 200 mg of preformed DHA per 92-gram sachet.
  Standard RUTF The standard RUTF used in the BrightSAM trial is a peanut butter paste with vegetable oil, skim milk powder, carbohydrates, vitamins, and minerals that is intended to cover the child's total daily nutritional needs. Standard RUTF will be manufactured in compliance with the specifications recommended by the Codex Alimentarius Commission17.
  Arms: eRUTF; sRUTF
Behavioral: Psychosocial stimulation — The psychosocial intervention has been developed and piloted for this study as a context-relevant adaptation from the WHO/UNICEF Care for Child Development package. It will be delivered in group sessions, where the primary caregiver will attend along with the child participating in the trial.
  During seven sessions of approximately two hours, caregivers will be trained on a variety of subjects which include; the first four sessions will be introductory and provide the basics of nutrition, the basics of psychosocial stimulation, and play and communication practices. We will build on the increasing experience of the caregivers and provide a deeper understanding of early child development.
  Standard nutritional counseling will adhere to national guidelines for pediatric management of severe acute malnutrition including nutritional counseling and psychosocial stimulation.
  Arms: PS; sNC

SUMMARY:
This is a randomized clinical trial to learn whether ready-to-use therapeutic foods enriched with choline and docosahexaenoic acid (DHA) together with psychosocial stimulating activities work well to improve child development in children with severe acute malnutrition(SAM). The overall question this trial aims to answer is can the health and development outcomes of children with SAM be improved through optimized nutritional treatment and integrated psychosocial support.

Researchers will compare the new ready-to-use therapeutic food and an integrated psychosocial stimulation to a standard look-alike nutritional supplement that contains no additional nutrients being investigated and the standard nutritional counseling given locally and assess its effects on child development in children with severe acute malnutrition.

Participants will:

* Be given the trial interventions which will be delivered over 12 weeks
* After the 12 weeks of intervention, participants will return for outcome evaluations (week 12 study visit), which will be repeated at follow-up visits after 24 and 48 weeks.

DETAILED DESCRIPTION:
Background Estimated, 13.6 million children were affected by severe acute malnutrition (SAM) in 2022. Early childhood is a critical period of brain development and children exposed to malnutrition in early life have poorer school performance and lower income in adult life. Introduction of Ready to use therapeutic foods (RUTF) has greatly improved the nutritional recovery of children with SAM. However, SAM remains associated with adverse effects on child cognitive and social development. The balance in the RUTF between polyunsaturated n-6 and n-3 essential fatty acids (EFAs) in RUTF has been questioned. Essential fatty acid (EFA) status is associated with child development, and children given the standard RUTF do not improve their n-3 EFA status after recovery.

A trial in Malawi found a positive effect on cognitive scores six months after completing nutritional therapy with RUTF with added preformed docosahexaenoic acid (DHA), a long-chain polyunsaturated fatty acid (PUFA) of the n-3 series, which is essential for neural growth. There is also a potential for improving the content of other nutrients of importance for neurodevelopment in early childhood like choline, which is essential for neurotransmitter synthesis and phospholipids in the brain. Studies have indicated a synergistic relationship between n-3 EFAs and choline, suggesting that low levels of one or both may negatively impact cognition.

Deficits in child development associated with SAM are not only caused by inadequate diets. Families exposed to malnutrition are often affected by psychological distress, consequently children are likely to be offered little stimulation and responsive care. However, in practice, support for psychosocial stimulation and responsive caregiving is rarely offered during hospital-based treatment, and it is still not included in the guidelines for community-based treatment of SAM. The intensity of this intervention is difficult under the constraints of most health services in low- and middle-income countries (LMIC). More recent packages for promoting responsive care have shown some effects, but often not when implemented at scale or within systems of care.

In this study we hypothesize that optimized nutritional treatment and integrated psychosocial support can improve the health and development outcomes of children with SAM.

Specific objectives:

1. to assess the effects of a modified RUTF and psychosocial stimulation, individually and combined, on attention, cognitive, motor, language and psycho-emotional development in children treated for SAM;
2. to investigate the pathways of intervention effects on cognitive development by assessing the role of DHA and choline status in the child as well as caregiver factors which include caregiver-child interaction, home stimulation and maternal psychological distress;
3. to assess how, why and for whom the modified RUTF and psychosocial interventions work within the trial context, perceptions of their feasibility of implementation within the routine health system, and the climate and environmental sustainability of interventions.

Methods:

This trial is designed as a 2x2 factorial randomized clinical trial to assess the effects of DHA and choline enriched vs. standard RUTF and psychosocial stimulation vs. standard counselling in management of SAM. Participants will be individually randomised to nutritional intervention arms and clusters will be randomized to psychosocial intervention arms.

The interventions will be delivered over a period of 12 weeks. After enrolment and baseline data collection, participants will receive their first RUTF sachets. They will then be requested to return to the study site for a total of seven visits during the intervention period to receive interventions. After the 12 weeks of intervention, participants will return for outcome evaluations (week 12 study visit), which will be repeated at follow-up visits after 24 and 48 weeks. The study will take place in Mwanza region, Tanzania. The trial will include children with uncomplicated SAM aged 6-36 months from eight health care facilities in Ilemela municipality, Nyamagana municipality and Magu district.

Outcomes:

The primary outcomes is the change in child development scores, which will be assessed at baseline, 12, 24 and 48 weeks and compared with intervention groups. These will assess gross, fine motor, language and psycho -emotional skills by validated tool called (MDAT) Malawi Development Assessment Tool) and neurocognitive function will be accessed by eye-tracking. Secondary outcomes will allow us to assess proximate effects of the interventions, which may mediate long-term effects on development

Analysis:

The primary analysis will be based on the intention-to-treat principle using available case data. The analysis will assess intervention effects based on the 2x2 factorial design by comparing changes in outcomes between baseline and intervention endline (i.e., 12 weeks) using a linear regression model adjusted for sex, age and month of inclusion to account for possible seasonal effects.

Secondary analysis will include assessment of intervention effects at 24- and 48-weeks follow-up using a linear mixed model to include repeated measurements. The models will include the baseline value of the outcome as fixed effect and participant as random effect to account for the correlation between measurements from the same participant. These models will also include adjustment for other variables as appropriate.

Secondary analyses will include per-protocol analyses to assess effects within groups with high compliance with the interventions

Ethics:

Ethical approval has been sought from the Medical Research Coordinating Committee (MRCC) of the National Institute for Medical Research in Tanzania and the London School of Hygiene and Tropical Medicine ethics committee.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 6-36 months.
2. Consent given by a caregiver older than 18 years.
3. Diagnosed with severe acute malnutrition (MUAC<115 mm, or WHZ ≤-3 or bipedal pitting edema).
4. Eligible for RUTF treatment (expanded below).

Exclusion Criteria:

1. Conditions preventing the child from receiving interventions, e.g., peanut butter allergy or cleft palate.
2. Moderate or severe disability which significantly affects normal child development (e.g., cerebral palsy or hydrocephalus), identified using a standardized screening form.
3. Children of families not living in the area or planning to move from the area within the follow-up period

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2025-11-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Change in MDAT scores | Assessed at baseline, 12, 24 and 48 weeks
  Development will be assessed by validated methods and include:
  Gross motor, fine motor, language, and psycho-emotional skills assessed by the Malawi Development assessment tool (MDAT)
Change in eye tracking scores | Baseline, 12, 24 and 48 weeks
  Neurocognitive function assessed by eye-tracking technique

SECONDARY OUTCOMES:
Level of caregiver stimulation and support | Assessed at baseline, 12, 24 and 48 weeks
  Caregiver stimulation and support assessed by Observations of Mother and Child Interactions (OMCI) questionnaire
Fatty acid composition | at baseline and at week 12, and week 48
  - Fatty acid composition assessed by gas chromatography
Mid upper arm circumference (MUAC) | Baseline, weekly, 12, 24 and 48 weeks
  - MUAC assessed using non-stretchable tape measure
Mortality | 12, 24 and 48 weeks
  Proportion of children who die during follow-up
Process evaluation | Interviews will be conducted after the last PS session ( Week 11) , and where possible, again with the same caregivers at long term follow-up (week 24 and 48).
  The process evaluation will examine the following aspects of the interventions:
  * Implementation
  * Mechanisms
  * Context
  * Acceptability
  * Feasibility of implementation within the health system
  * Programme theory
Levels of choline | Baseline, 12, 24 and 48 weeks
  Levels of choline and related metabolites assessed by mass spectrometry
C-reactive protein (CRP) | Baseline, 12, 24 and 48 weeks
  Serum CRP assessed as a marker of systemic inflammation
Ferritin | Baseline, 12, 24 and 48 weeks
  Serum ferritin assessed as marker of iron status
Level of Alanine transaminase | Baseline, 12, 24 and 48 weeks
  Serum alanine transaminase as a marker of liver function
Level of Aspartate transaminase | Baseline, 12, 24 and 48 weeks
  Serum aspartate transaminase assessed as a marker of liver function
Level of maternal psychological distress | Baseline, 12, 24 and 48 weeks
  Maternal psychological distress assessed by Patient Health Questionnaire 9 (PHQ-9)
Status of the learning environment | Baseline, 12, 24 and 48 weeks
  The status of learning environment assessed by the Family Care Indicators (FCI) questionnaire
Status of maternal social support framework | Baseline, 12, 24 and 48 weeks
  The status of maternal social support framework assessed by the Multidimensional Scale of Perceived Social Support questionnaire
Morbidity | 12, 24 and 48 weeks
  . Proportion of children with one or multiple illness episodes during follow-up
- Weight-for-height z-score (WHZ) | Baseline, 12, 24 and 48 weeks
  - Weight-for-height z-score (WHZ) based on length/height (m) and weight (kg) measurements'
Height-for-age z-score (HAZ) , based on length/height and age) | Baseline, 12, 24 and 48 weeks
  Height-for-age z-score (HAZ) assessed based on length/height (m) and age (month)
Rate of nutritional recovery at the end of intervention period | 12
  Rate of nutritional recovery at the end of intervention period, defined as WHZ > -2 and MUAC > 125 mm, and no bilateral pitting oedema for two weeks
Proportion relapsing to moderate acute malnutrition (MAM) after recovery | 12 weeks
  Proportion relapsing to moderate acute malnutrition (MAM) after recovery, measured as WHZ ≤ -2 and >-3 or MUAC ≤ 125 and >115mm)
Proportion relapsing to SAM after recovery | Any time point, 24 and 48 weeks
  Proportion relapsing to SAM after recovery, measured as WHZ <-3, MUAC <115mm or presence of nutritional oedema, assessed at any caregiver-initiated contacts to the study site at any point during the 48 weeks of follow-up and at study visits at 24 and 48 weeks
Implementation evaluation | Interviews will be conducted after the last PS session ( Week 11) , and where possible, again with the same caregivers at long term follow-up (week 24 and 48).
  The implementation component will assess
  * The fidelity of implementation of each component of the intervention,
  * The dose (amount, frequency) of each component delivered to the children,
  * Any adaptations to the intervention and why these were made,
  * The reach of the interventions, provider and caregiver experience
  * Perceptions, mechanisms and any unintended consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Olsen, MSc, PhD, Principal Investigator — Rigshospitalet, Denmark; George PrayGod, MD, PhD, Principal Investigator — National Institute for Medical Research
Locations (1):
- National Institute for Medical Research, Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grantham-McGregor S, Stewart ME, Schofield WN. Effect of long-term psychosocial stimulation on mental development of severely malnourished children. Lancet. 1980 Oct 11;2(8198):785-9. doi: 10.1016/s0140-6736(80)90395-5. PMID 6107460
- [Background] Olsen MF, Iuel-Brockdorff AS, Yameogo CW, Cichon B, Fabiansen C, Filteau S, Phelan K, Ouedraogo A, Wells JC, Briend A, Michaelsen KF, Lauritzen L, Ritz C, Ashorn P, Christensen VB, Gladstone M, Friis H. Early development in children with moderate acute malnutrition: A cross-sectional study in Burkina Faso. Matern Child Nutr. 2020 Apr;16(2):e12928. doi: 10.1111/mcn.12928. Epub 2019 Dec 11. PMID 31823490
- [Background] Stephenson K, Callaghan-Gillespie M, Maleta K, Nkhoma M, George M, Park HG, Lee R, Humphries-Cuff I, Lacombe RJS, Wegner DR, Canfield RL, Brenna JT, Manary MJ. Low linoleic acid foods with added DHA given to Malawian children with severe acute malnutrition improve cognition: a randomized, triple-blinded, controlled clinical trial. Am J Clin Nutr. 2022 May 1;115(5):1322-1333. doi: 10.1093/ajcn/nqab363. PMID 34726694
- [Background] Gera T, Pena-Rosas JP, Boy-Mena E, Sachdev HS. Lipid based nutrient supplements (LNS) for treatment of children (6 months to 59 months) with moderate acute malnutrition (MAM): A systematic review. PLoS One. 2017 Sep 21;12(9):e0182096. doi: 10.1371/journal.pone.0182096. eCollection 2017. PMID 28934235
- [Background] Lelijveld N, Jalloh AA, Kampondeni SD, Seal A, Wells JC, Goyheneix M, Chimwezi E, Mallewa M, Nyirenda MJ, Heyderman RS, Kerac M. Brain MRI and cognitive function seven years after surviving an episode of severe acute malnutrition in a cohort of Malawian children. Public Health Nutr. 2019 Jun;22(8):1406-1414. doi: 10.1017/S1368980018003282. Epub 2018 Dec 3. PMID 30501662
- [Background] Hoddinott J, Behrman JR, Maluccio JA, Melgar P, Quisumbing AR, Ramirez-Zea M, Stein AD, Yount KM, Martorell R. Adult consequences of growth failure in early childhood. Am J Clin Nutr. 2013 Nov;98(5):1170-8. doi: 10.3945/ajcn.113.064584. Epub 2013 Sep 4. PMID 24004889
- See also: Levels and trends in child malnutrition: UNICEF/WHO/World Bank Group joint child malnutrition estimates: key findings of the 2023 edition — https://www.who.int/publications/i/item/9789240073791